CLINICAL TRIAL: NCT00655954
Title: Osteoprotegerin (OPG) in Induced Sputum as a Novel Biomarker for COPD
Brief Title: Osteoprotegerin (OPG) in Induced Chronic Obstructive Pulmonary Disease (COPD) Sputum
Status: Completed | Type: Observational
Sponsor: Imperial College London (Other)
Responsible Party: Sponsor
Other Study IDs: 05-Q0407-91
Record Dates: First submitted 2008-04-04; First posted 2008-04-10 (Estimated); Last update posted 2019-07-10 (Actual); Status verified 2019-07

CONDITIONS: Pulmonary Disease, Chronic Obstructive
Keywords: COPD; asthma; smokers; healthy volunteers; bronchiectasis; cystic fibrosis
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Asthma; Bronchiectasis; Cystic Fibrosis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Healthy volunteers non smoker: 18 volunteers
  Interventions: Procedure: Induced sputum
- Healthy volunteers smoker: 15 volunteers
  Interventions: Procedure: Induced sputum
- Chronic Obstructive Pulmonary Disease COPD: 39 volunteers
  Interventions: Procedure: Induced sputum

INTERVENTIONS:
Procedure: Induced sputum — Used Ultrasonic nebuliser

SUMMARY:
Evaluation of OPG level as disease markers has also been reported. It has been showed that patients with coronary artery disease had higher serum OPG levels than healthy volunteers. Moreover, serum OPG levels correlate with the number of stenotic coronary arteries

DETAILED DESCRIPTION:
Osteoprotegerin (OPG) is a secreted glycoprotein containing 401 amino acids. It is a member of the tumour necrosis factor (TNF) receptor superfamily. It was firstly discovered as a protein regulating bone metabolism, inhibiting osteoclastogenesis, consequently, inhibiting bone resorption OPG is detected in lung using Northern blot analysis. It is likely that OPG would contribute to the pathogenesis of COPD and could be an effective disease marker of the disease

ELIGIBILITY:
Inclusion Criteria:

* Healthy non-smokers

  * Age <35 years (younger group)
  * Aged matched to COPD patients (older group)
  * Normal spirometry
  * Subjects are able to give informed consent
* Healthy smokers

  * Age <35 years (younger group)
  * Aged matched to COPD patients (older group)
  * Normal spirometry
  * Subjects are able to give informed consent Stable COPD patients: Stage I-IV according to the GOLD guidelines (3), (9)
  * Current and/or ex-smokers with no less than 10 pack-year smoking history
  * The subjects are able to give informed consent COPD patients with acute exacerbation: Stage I-IV according to the GOLD guidelines (3), (9)
  * Exacerbation of COPD defined as "an event in the natural course of the disease characterised by a change in the patient's baseline dyspnoea, cough and/or sputum beyond day to day variability sufficient to warrant a change in management" (9)
  * Current and/or ex-smokers with no less than 10 pack-year smoking history
  * The subjects are able to give informed consent Asthma patients
  * Patients diagnosed with asthma
  * The subjects are able to give informed consent Bronchiectasis patients
  * Patients with CT-confirmed bronchiectasis
  * The subjects are able to give informed consent Cystic fibrosis patients
  * Patients diagnosed with cystic fibrosis
  * The subjects are able to give informed consent

Exclusion Criteria:

* Healthy non-smokers and smokers

  * Upper respiratory infection within the last 4 weeks.
  * Subjects who have received research medication within the previous one month.
  * Subjects unable to give informed consent.
  * Any psychiatric condition rendering the patient unable to understand the nature, scope and possible consequences of the study Stable COPD patients
  * Patients who have had an exacerbation which required treatment with oral steroids during the last 2 months prior to the visit
  * Upper respiratory infection within the last 4 weeks
  * Subjects who have received research medication within the previous one month
  * Subjects unable to give informed consent
  * Any psychiatric condition rendering the patient unable to understand the nature, scope and possible consequences of the study COPD patients with acute exacerbation
  * Subjects who have received research medication within the previous one month
  * Subjects unable to give informed consent
  * Any psychiatric condition rendering the patient unable to understand the nature, scope and possible consequences of the study Asthma
  * Upper respiratory infection within the last 4 weeks
  * Subjects who have received research medication within the previous one month
  * Subjects unable to give informed consent.
  * Any psychiatric condition rendering the patient unable to understand the nature, scope and possible consequences of the study.
* Bronchiectasis and cystic fibrosis

  * Subjects who have received research medication within the previous one month.
  * Subjects unable to give informed consent.
  * Any psychiatric condition rendering the patient unable to understand the nature, scope and possible consequences of the study.

Min Age: 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants were recruited from the outpatient department of Royal Brompton Hospital and local general practices. Patients with COPD were diagnosed using the GOLD (Global Initiative for Obstructive Lung Disease) criteria. 25 Patients with COPD who had an exacerbation during the last 2 months prior to the visit were excluded. Patients with asthma were diagnosed using the GINA (Global Initiative for Asthma) guidelines for asthma. 26 Patients with any other lung diseases were excluded from the study. This study was reviewed and approved by the Hounslow and Hillingdon Research Ethics Committee. Written informed consent was obtained from all subjects.
Sampling Method: Non-Probability Sample
Enrollment: 72 (Actual)
Dates: Start 2008-01 (Actual); Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
Sputum OPG | 1 hour
  Sputum OPG as assessed by ELISA at baseline

CONTACTS AND LOCATIONS:
Overall Officials: Sergei A Kharitonov, MD PhD, Principal Investigator — National Heart and Lung Institute
Locations (1):
- National Heart and Lung Institute, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] To M, Ito K, Ausin PM, Kharitonov SA, Barnes PJ. Osteoprotegerin in sputum is a potential biomarker in COPD. Chest. 2011 Jul;140(1):76-83. doi: 10.1378/chest.10-1608. Epub 2010 Dec 2. PMID 21127170